CLINICAL TRIAL: NCT03214250
Title: Open-label, Multicenter, Phase 1b/2 Clinical Study to Evaluate the Safety and Efficacy of CD40 Agonistic Monoclonal Antibody (APX005M) Administered Together With Gemcitabine and Nab-Paclitaxel With or Without PD-1 Blocking Antibody (Nivolumab) in Patients With Previously Untreated Metastatic Pancreatic Adenocarcinoma
Brief Title: Safety and Efficacy of APX005M With Gemcitabine and Nab-Paclitaxel With or Without Nivolumab in Patients With Previously Untreated Metastatic Pancreatic Adenocarcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Parker Institute for Cancer Immunotherapy (Other)
Collaborators: Bristol-Myers Squibb (Industry); Apexigen America, Inc. (Industry); Cancer Research Institute, New York City (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PICI0002; UPCC 11217 (Other: University of Pennsylvania)
Record Dates: First submitted 2017-06-09; First posted 2017-07-11 (Actual); Results first posted 2022-08-11 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Metastatic Pancreatic Adenocarcinoma
Keywords: Nivolumab; APX005M; previously untreated metastatic pancreatic adenocarcinoma; Gemcitabine; nab-Paclitaxel
MeSH Terms: interventions — sotigalimab; Nivolumab; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Gem/NP/nivolumab (Experimental): Gemcitabine+Nab-Paclitaxel+nivolumab
  Interventions: Drug: Nivolumab; Drug: Nab-Paclitaxel; Drug: Gemcitabine
- Gem/NP/APX005M (Experimental): Gemcitabine+Nab-Paclitaxel+APX005M
  Interventions: Drug: APX005M; Drug: Nab-Paclitaxel; Drug: Gemcitabine
- Gem/NP/nivolumab/APX005M (Experimental): Gemcitabine+Nab-Paclitaxel+nivolumab+APX005M
  Interventions: Drug: APX005M; Drug: Nivolumab; Drug: Nab-Paclitaxel; Drug: Gemcitabine

INTERVENTIONS:
Drug: APX005M — Administer intravenously once every 28-day Cycle
  Arms: Gem/NP/APX005M; Gem/NP/nivolumab/APX005M
Drug: Nivolumab — Administer intravenously twice every 28-day cycle
  Other Names: Opdivo
  Arms: Gem/NP/nivolumab; Gem/NP/nivolumab/APX005M
Drug: Nab-Paclitaxel — Administer intravenously on 3 times every 28-day cycle
  Other Names: Abraxane
Drug: Gemcitabine — Administer intravenously 3 times every 28-day cycle
  Other Names: Gemzar

SUMMARY:
The main purposes of this study are to learn how effective the study drug combinations are in treating patients with metastatic pancreatic adenocarcinoma. The drug combinations are APX005M+Nivolumab+Gemcitabine+nab-Paclitaxel, or APX005M+Gemcitabine+nab-Paclitaxel.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has histologically or cytologically documented diagnosis of pancreatic adenocarcinoma with metastatic disease. Locally advanced subjects are not eligible.
2. Subject must have measureable disease by RECIST 1.1.
3. Subjects must be age 18 years or older.
4. Subjects must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
5. Subjects must have the following laboratory values at screening within 2 weeks of the first dose of investigational agents:

   * Absolute neutrophil count (ANC) ≥1.5 x 109/L (in absence of growth factor support)
   * Platelet count ≥150 x 109/L
   * Hemoglobin ≥9 g/dL(without transfusion support)
   * Serum creatinine ≤1.5 mg/dL, and creatinine clearance ≥ 50 ml/min as measured by Cockcroft and Gault formula
   * Aspartate aminotransferase (AST) and ALT ≤2.5 x upper limit of normal (ULN)
   * Total bilirubin ≤1.5 x ULN, except in subjects with documented Gilbert's Syndrome, who must have a total bilirubin ≤3 x ULN
6. Women of childbearing potential (WOCBP) must have a negative pregnancy test (serum or urine) within the 7 days prior to study drug administration, and within the 3 days before the first study drug administration, or a negative pregnancy test within the 24 hours before the first study drug administration.
7. WOCBP and male subjects who are sexually active with WOCBP must agree to use 2 highly effective methods of contraception (including a physical barrier) before the first dose of study drugs, during the study, and for 5 months for women and 7 months for men following the last dose of study drug.
8. Subjects must have the ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

1. Subject must not have received any prior treatment, including chemotherapy, biological therapy, or targeted therapy for metastatic pancreatic adenocarcinoma, with the following exceptions and notes:

   1. Subjects who have received prior adjuvant therapy for pancreatic adenocarcinoma are eligible if neoadjuvant and adjuvant therapy (including chemotherapy and/or radiotherapy) was fully completed more than 4 months before the start of study treatment. In this case, prior Gem and/or NP is allowable
   2. Prior resection surgery is allowable.
   3. Patients initially diagnosed with locally advanced pancreatic cancer who have undergone chemotherapy then resection and were with no evidence of disease are eligible if metastatic relapse of disease has occurred and if the last dose of chemotherapy was more than 4 months before the data of study entry.
2. Subjects must not have another active invasive malignancy, with the following exceptions and notes:

   1. History of a non-invasive malignancy, such as cervical cancer in situ, non-melanomatous carcinoma of the skin, in situ melanoma, or ductal carcinoma in situ of the breast, is allowed.
   2. History of malignancy that is in complete remission after treatment with curative intent is allowed.
   3. No current or history of a hematologic malignancy is allowed, including subjects who have undergone a bone marrow transplant.
3. History of clinically significant sensitivity or allergy to monoclonal antibodies, their excipients, or intravenous gamma globulin
4. Previous exposure to CD40, PD-1, PD-L1, CTLA-4 antibodies or any other immunomodulatory agent
5. History of (non-infectious) pneumonitis that required corticosteroids or current pneumonitis, or history of interstitial lung disease
6. Subjects must not have a known or suspected history of an autoimmune disorder, including but not limited to inflammatory bowel disease, celiac disease, Wegner syndrome, Hashimoto syndrome, systemic lupus erythematosus, scleroderma, sarcoidosis, or autoimmune hepatitis, within 3 years of the first dose of investigational agent, except for the following.

   a. Subjects with Type 1 diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders such as vitiligo, or alopecia not requiring systemic therapy, or conditions not expected to recur in the absence of an external trigger are eligible.
7. Subjects must not have an uncontrolled intercurrent illness, including an ongoing or active infection, current pneumonitis, symptomatic congestive heart failure (New York Heart Association class III or IV), unstable angina, uncontrolled hypertension, cardiac arrhythmia, interstitial lung disease, active coagulopathy, or uncontrolled diabetes.
8. Subjects must not have a history of myocardial infarction within 6 months or a history of arterial thromboembolic event within 3 months of the first dose of investigational agent.
9. Subjects must not have a history of human immunodeficiency virus, hepatitis B, or hepatitis C, except for the following:

   1. subjects with anti-hepatitis B core antibody but with undetectable HBV DNA and negative for HBsAg
   2. subjects with resolved or treated HCV (i.e. HCV antibody positive but undetectable HCV RNA)
10. Subjects must not have a history of primary immunodeficiency.
11. Subjects must not receive concurrent or prior use of an immunosuppressive agent within 14 days of the first dose of investigational agent, with the following exceptions and notes:

    1. Systemic steroids at physiologic doses (equivalent to dose of oral prednisone 10 mg) are permitted. Steroids as anti-emetics for chemotherapy are not allowed.
    2. Intranasal, inhaled, topical, intra-articular, and ocular corticosteroids with minimal systemic absorption are permitted.
    3. Subjects with a condition with anticipated use of systemic steroids above the equivalent of 10 mg prednisone are excluded.
12. Subjects must not have a history of clinically manifested central nervous system (CNS) metastases.

    a. Subjects with known or suspected leptomeningeal disease or cord compression are not eligible.
13. Subjects must not have had major surgery as determined by the PI within 4 weeks before the first dose of investigational agent.
14. Subjects must not have received another investigational agent within the shorter of 4 weeks or 5 half-lives before the first dose of investigational agent.
15. Subjects must not have received a live attenuated vaccine within 28 days before the first dose of investigational agent, and subjects, if enrolled, should not receive live vaccines during the study or for 180 days after the last dose of investigational agent.
16. Females who are pregnant or lactating or who intend to become pregnant during participation in the study are not eligible to participate.
17. Subjects who are of reproductive potential who refuse to use effective methods of birth control during the course of participation of the study and within 5 month for women and 7 months for men of the last dose of investigational agent are ineligible to participate in the study.
18. Subjects who have any clinically significant psychiatric, social, or medical condition that, in the opinion of the investigator, could increase the subject's risk, interfere with protocol adherence, or affect the subject's ability to give informed consent are ineligible to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2017-07-21 (Actual); Primary Completion 2021-02-11 (Actual); Study Completion 2022-02-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Parker Institute for Cancer Immunotherapy, Study Director — Parker Institute for Cancer Immunotherapy
Locations (7):
- United States (7):
  - University of California, Los Angeles, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Stanford University, Stanford, California
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Pennsylvania, Abramson Cancer Center, Philadelphia, Pennsylvania
  - M.D. Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rahib L, Smith BD, Aizenberg R, Rosenzweig AB, Fleshman JM, Matrisian LM. Projecting cancer incidence and deaths to 2030: the unexpected burden of thyroid, liver, and pancreas cancers in the United States. Cancer Res. 2014 Jun 1;74(11):2913-21. doi: 10.1158/0008-5472.CAN-14-0155. PMID 24840647
- [Background] Von Hoff DD, Ervin T, Arena FP, Chiorean EG, Infante J, Moore M, Seay T, Tjulandin SA, Ma WW, Saleh MN, Harris M, Reni M, Dowden S, Laheru D, Bahary N, Ramanathan RK, Tabernero J, Hidalgo M, Goldstein D, Van Cutsem E, Wei X, Iglesias J, Renschler MF. Increased survival in pancreatic cancer with nab-paclitaxel plus gemcitabine. N Engl J Med. 2013 Oct 31;369(18):1691-703. doi: 10.1056/NEJMoa1304369. Epub 2013 Oct 16. PMID 24131140
- [Background] Pardoll DM. The blockade of immune checkpoints in cancer immunotherapy. Nat Rev Cancer. 2012 Mar 22;12(4):252-64. doi: 10.1038/nrc3239. PMID 22437870
- [Background] Bauer C, Kuhnemuth B, Duewell P, Ormanns S, Gress T, Schnurr M. Prevailing over T cell exhaustion: New developments in the immunotherapy of pancreatic cancer. Cancer Lett. 2016 Oct 10;381(1):259-68. doi: 10.1016/j.canlet.2016.02.057. Epub 2016 Mar 8. PMID 26968250
- [Background] Khong A, Nelson DJ, Nowak AK, Lake RA, Robinson BW. The use of agonistic anti-CD40 therapy in treatments for cancer. Int Rev Immunol. 2012 Aug;31(4):246-66. doi: 10.3109/08830185.2012.698338. PMID 22804570
- [Background] Topalian SL, Hodi FS, Brahmer JR, Gettinger SN, Smith DC, McDermott DF, Powderly JD, Carvajal RD, Sosman JA, Atkins MB, Leming PD, Spigel DR, Antonia SJ, Horn L, Drake CG, Pardoll DM, Chen L, Sharfman WH, Anders RA, Taube JM, McMiller TL, Xu H, Korman AJ, Jure-Kunkel M, Agrawal S, McDonald D, Kollia GD, Gupta A, Wigginton JM, Sznol M. Safety, activity, and immune correlates of anti-PD-1 antibody in cancer. N Engl J Med. 2012 Jun 28;366(26):2443-54. doi: 10.1056/NEJMoa1200690. Epub 2012 Jun 2. PMID 22658127
- [Derived] Padron LJ, Maurer DM, O'Hara MH, O'Reilly EM, Wolff RA, Wainberg ZA, Ko AH, Fisher G, Rahma O, Lyman JP, Cabanski CR, Yu JX, Pfeiffer SM, Spasic M, Xu J, Gherardini PF, Karakunnel J, Mick R, Alanio C, Byrne KT, Hollmann TJ, Moore JS, Jones DD, Tognetti M, Chen RO, Yang X, Salvador L, Wherry EJ, Dugan U, O'Donnell-Tormey J, Butterfield LH, Hubbard-Lucey VM, Ibrahim R, Fairchild J, Bucktrout S, LaVallee TM, Vonderheide RH. Sotigalimab and/or nivolumab with chemotherapy in first-line metastatic pancreatic cancer: clinical and immunologic analyses from the randomized phase 2 PRINCE trial. Nat Med. 2022 Jun;28(6):1167-1177. doi: 10.1038/s41591-022-01829-9. Epub 2022 Jun 3. PMID 35662283
- [Derived] O'Hara MH, O'Reilly EM, Varadhachary G, Wolff RA, Wainberg ZA, Ko AH, Fisher G, Rahma O, Lyman JP, Cabanski CR, Mick R, Gherardini PF, Kitch LJ, Xu J, Samuel T, Karakunnel J, Fairchild J, Bucktrout S, LaVallee TM, Selinsky C, Till JE, Carpenter EL, Alanio C, Byrne KT, Chen RO, Trifan OC, Dugan U, Horak C, Hubbard-Lucey VM, Wherry EJ, Ibrahim R, Vonderheide RH. CD40 agonistic monoclonal antibody APX005M (sotigalimab) and chemotherapy, with or without nivolumab, for the treatment of metastatic pancreatic adenocarcinoma: an open-label, multicentre, phase 1b study. Lancet Oncol. 2021 Jan;22(1):118-131. doi: 10.1016/S1470-2045(20)30532-5. PMID 33387490

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1b: Gem/NP/APX005M (0.1 mg/kg): Gemcitabine+Nab-Paclitaxel+APX005M (0.1 mg/kg)
  APX005M: Administer intravenously once every 28-day Cycle
  Nab-Paclitaxel: Administer intravenously on 3 times every 28-day cycle
  Gemcitabine: Administer intravenously 3 times every 28-day cycle
- Phase 1b: Gem/NP/APX005M (0.3 mg/kg); Phase 2: Gem/NP/APX005M (0.3 mg/kg): Gemcitabine+Nab-Paclitaxel+APX005M (0.3 mg/kg)
  APX005M: Administer intravenously once every 28-day Cycle
  Nab-Paclitaxel: Administer intravenously on 3 times every 28-day cycle
  Gemcitabine: Administer intravenously 3 times every 28-day cycle
- Phase 1b: Gem/NP/Nivolumab/APX005M (0.1 mg/kg): Gemcitabine+Nab-Paclitaxel+nivolumab+APX005M (0.1 mg/kg)
  APX005M: Administer intravenously once every 28-day Cycle
  Nivolumab: Administer intravenously twice every 28-day cycle
  Nab-Paclitaxel: Administer intravenously on 3 times every 28-day cycle
  Gemcitabine: Administer intravenously 3 times every 28-day cycle
- Phase 1b: Gem/NP/Nivolumab/APX005M (0.3 mg/kg); Phase 2: Gem/NP/Nivolumab/APX005M (0.3 mg/kg): Gemcitabine+Nab-Paclitaxel+nivolumab+APX005M (0.3 mg/kg)
  APX005M: Administer intravenously once every 28-day Cycle
  Nivolumab: Administer intravenously twice every 28-day cycle
  Nab-Paclitaxel: Administer intravenously on 3 times every 28-day cycle
  Gemcitabine: Administer intravenously 3 times every 28-day cycle
- Phase 2: Gem/NP/Nivolumab: Gemcitabine+Nab-Paclitaxel+nivolumab
  Nivolumab: Administer intravenously twice every 28-day cycle
  Nab-Paclitaxel: Administer intravenously on 3 times every 28-day cycle
  Gemcitabine: Administer intravenously 3 times every 28-day cycle
Period: Overall Study
Arm/Group | Phase 1b: Gem/NP/APX005M (0.1 mg/kg) | Phase 1b: Gem/NP/APX005M (0.3 mg/kg) | Phase 1b: Gem/NP/Nivolumab/APX005M (0.1 mg/kg) | Phase 1b: Gem/NP/Nivolumab/APX005M (0.3 mg/kg) | Phase 2: Gem/NP/Nivolumab | Phase 2: Gem/NP/APX005M (0.3 mg/kg) | Phase 2: Gem/NP/Nivolumab/APX005M (0.3 mg/kg)
Started | 7 | 7 | 8 | 8 | 37 | 31 | 31
Completed (Per the protocol, "completed" status is defined as completing 5 years of survival follow-up from the time a patient has discontinued treatment.) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 7 | 7 | 8 | 8 | 37 | 31 | 31
Not completed — Death | 5 | 5 | 7 | 4 | 23 | 23 | 24
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 1 | 2 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 1 | 1 | 2
Not completed — Remains on Study | 2 | 2 | 0 | 1 | 7 | 5 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 2 | 5 | 0 | 2

BASELINE CHARACTERISTICS:
Population: The Phase 1b Safety Population is defined as all patients who were enrolled in Phase 1b and who received at least 1 dose of any study drug. The Phase 2 Efficacy Population is defined as all patients who were randomized in Phase 2 and who received at least 1 dose of any study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1b: Gem/NP/APX005M (0.1 mg/kg) | Phase 1b: Gem/NP/APX005M (0.3 mg/kg) | Phase 1b: Gem/NP/Nivolumab/APX005M (0.1 mg/kg) | Phase 1b: Gem/NP/Nivolumab/APX005M (0.3 mg/kg) | Phase 2: Gem/NP/Nivolumab | Phase 2: Gem/NP/APX005M (0.3 mg/kg) | Phase 2: Gem/NP/Nivolumab/APX005M (0.3 mg/kg) | Total
Number analyzed (Participants) | 7 | 7 | 8 | 8 | 37 | 31 | 31 | 129
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 4 | 1 | 6 | 21 | 18 | 18 | 70
  >=65 years | 5 | 3 | 7 | 2 | 16 | 13 | 13 | 59
Age, Continuous [Median (Full Range); unit: years] | 66.0 [52 to 73] | 64.0 [54 to 76] | 70.0 [61 to 79] | 61.0 [39 to 71] | 64.0 [47 to 75] | 60.0 [35 to 78] | 62 [34 to 78] | 63.0 [34 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 3 | 4 | 16 | 11 | 13 | 54
  Male | 2 | 5 | 5 | 4 | 21 | 20 | 18 | 75
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 4
  Not Hispanic or Latino | 7 | 7 | 8 | 8 | 36 | 30 | 29 | 125
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 0 | 0 | 1 | 1 | 3 | 4 | 1 | 10
  Race: Black or African American | 0 | 1 | 0 | 1 | 0 | 2 | 1 | 5
  Race: White | 7 | 6 | 7 | 6 | 32 | 24 | 26 | 108
  Race: Other | 0 | 0 | 0 | 0 | 2 | 1 | 3 | 6
ECOG Performance Score [Count of Participants; unit: Participants] — The Eastern Cooperative Oncology Group (ECOG) Scale of Performance Status is one such measurement. It describes a patient's level of functioning in terms of their ability to care for themself, daily activity, and physical ability (walking, working, etc.). The ECOG Performance Status ranges from 0 (fully active, able to carry on all pre-disease performance without restriction) to 5 (dead).
  Participants
    ECOG Score = 0 | 3 | 1 | 5 | 4 | 17 | 19 | 14 | 63
    ECOG Score = 1 | 4 | 6 | 3 | 4 | 20 | 12 | 17 | 66
Cancer Location [Count of Participants; unit: Participants]
  Pancreas Body | 2 | 4 | 4 | 1 | 13 | 6 | 9 | 39
  Pancreas Head | 4 | 3 | 2 | 6 | 15 | 15 | 15 | 60
  Pancreas Tail | 1 | 0 | 2 | 1 | 9 | 10 | 7 | 30
Prior Treatment [Count of Participants; unit: Participants]
  Prior Chemotherapy: Yes | 3 | 2 | 1 | 3 | 9 | 5 | 4 | 27
  Prior Chemotherapy: No | 4 | 5 | 7 | 5 | 28 | 26 | 27 | 102
  Prior Cancer Surgery: Yes | 3 | 3 | 1 | 4 | 11 | 8 | 5 | 35
  Prior Cancer Surgery: No | 4 | 4 | 7 | 4 | 26 | 23 | 26 | 94
  Prior Radiation: Yes | 1 | 0 | 1 | 3 | 7 | 1 | 2 | 15
  Prior Radiation: No | 6 | 7 | 7 | 5 | 30 | 30 | 29 | 114
Cancer Stage at Initial Diagnosis [Count of Participants; unit: Participants]
  Stage 1 | 0 | 1 | 0 | 0 | 0 | 0 | 4 | 5
  Stage 2 | 2 | 3 | 2 | 4 | 4 | 4 | 2 | 21
  Stage 3 | 1 | 0 | 0 | 0 | 3 | 1 | 1 | 6
  Stage 4 | 4 | 3 | 6 | 4 | 30 | 26 | 24 | 97

OUTCOME MEASURES:

1. Primary Outcome: Phase 1b Primary Safety Outcome
Description: Number and percentage of subjects with adverse events (AEs), serious adverse events (SAEs), and dose-limiting toxicities (DLTs)
Time Frame: Initiation of study drug (or informed consent for SAEs) through 100 days after the last dose of study drug or initiation of a new systemic anti-cancer therapy with a maximum exposure of 34.3 months.
Population: The DLT-Evaluable Population is defined as all Phase 1b patients who received at least 2 doses of NP, at least 2 doses of Gem, and 1 dose of APX005M during Cycle 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: Gem/NP/APX005M (0.1 mg/kg) | Phase 1b: Gem/NP/APX005M (0.3 mg/kg) | Phase 1b: Gem/NP/Nivolumab/APX005M (0.1 mg/kg) | Phase 1b: Gem/NP/Nivolumab/APX005M (0.3 mg/kg)
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants
  Adverse Events (AEs) | 6 | 6 | 6 | 6
  Serious Adverse Events (SAEs) | 4 | 4 | 6 | 1
  Dose-Limiting Toxicities (DLTs) | 0 | 1 | 1 | 0

2. Primary Outcome: 1-year Overall Survival Rate
Description: The primary endpoint was the 1-year OS rate of each treatment arm, compared to the historical rate of 35% for gemcitabine and nab-Paclitaxel. OS was defined as the time from treatment initiation until death from any cause. Patients who were not reported as having died at the time of analysis were censored at the most recent contact date. OS and the 1-year OS rate were estimated by the Kaplan-Meier method for each treatment arm. The 1-year OS rate and corresponding one-sided, 95% CI were calculated to determine whether the lower bound of the CI excluded the assumed historical value of 35%. P values were calculated using a one-sided, one-sample z-test of the Kaplan-Meier estimate of the 1-year OS rate (and its standard error) against the historical rate of 35%. This study was not powered for statistical comparison between arms.
Time Frame: 1 year from initiation of study therapy
Population: The Efficacy Population is defined as (1) all patients who were randomized in Phase 2 and who received at least 1 dose of any study drug and (2) the 12 DLT-evaluable patients enrolled in Phase 1b at the recommended Phase 2 dose.
Measure: Number (95% Confidence Interval); unit: probability
Groups:
- Gem/NP/APX005M (0.3 mg/kg): Gemcitabine+Nab-Paclitaxel+APX005M (0.3 mg/kg)
  APX005M: Administer intravenously once every 28-day Cycle
  Nab-Paclitaxel: Administer intravenously on 3 times every 28-day cycle
  Gemcitabine: Administer intravenously 3 times every 28-day cycle
- Gem/NP/Nivolumab/APX005M (0.3 mg/kg): Gemcitabine+Nab-Paclitaxel+nivolumab+APX005M (0.3 mg/kg)
  APX005M: Administer intravenously once every 28-day Cycle
  Nivolumab: Administer intravenously twice every 28-day cycle
  Nab-Paclitaxel: Administer intravenously on 3 times every 28-day cycle
  Gemcitabine: Administer intravenously 3 times every 28-day cycle
Arm/Group | Gem/NP/Nivolumab | Gem/NP/APX005M (0.3 mg/kg) | Gem/NP/Nivolumab/APX005M (0.3 mg/kg)
Number analyzed (Participants) | 34 | 36 | 35
probability | 0.577 [0.384 to 0.729] | 0.481 [0.309 to 0.634] | 0.413 [0.244 to 0.575]
Statistical Analysis 1: Comparison: Gem/NP/Nivolumab; Each treatment arm was analyzed independently and compared to a historical 1-year OS reference rate of 35%; Test type: Superiority — One-sided; p = 0.006, z-test — one-sided p-value; One-sided, one-sample z-test of the Kaplan-Meier estimate of the 1-year OS rate (and its standard error) against the historical rate of 35%; probability = 0.577, 95% CI 1-sided [lower limit 0.417]
Statistical Analysis 2: Comparison: Gem/NP/APX005M (0.3 mg/kg); Each treatment arm was analyzed independently and compared to a historical 1-year OS reference rate of 35%; Test type: Superiority — One-sided; p = 0.062, z-test — one-sided p-value; [statistical method as in outcome 2, analysis 1]; probability = 0.481, 95% CI 1-sided [lower limit 0.337]
Statistical Analysis 3: Comparison: Gem/NP/Nivolumab/APX005M (0.3 mg/kg); Each treatment arm was analyzed independently and compared to a historical 1-year OS reference rate of 35%; Test type: Superiority — One-sided; p = 0.233, z-test — one-sided p-value; [statistical method as in outcome 2, analysis 1]; probability = 0.413, 95% CI 1-sided [lower limit 0.270]

3. Secondary Outcome: Objective Response Rate (ORR): DLT-Evaluable Population
Description: Phase 1b DLT-Evaluable Population. Overall Response Rate is defined as the proportion of participants who had a best overall response of Complete Response (CR) or Partial Response (PR) as defined by RECIST v1.1. Overall Response (OR) = CR + PR.
Time Frame: Initiation of study drug through radiographic progression or initiation of new anti-cancer therapy with a maximum exposure of 34.3 months.
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Gem/NP/APX005M (0.1 mg/kg): Gemcitabine+Nab-Paclitaxel+APX005M (0.1 mg/kg)
  APX005M: Administer intravenously once every 28-day Cycle
  Nab-Paclitaxel: Administer intravenously on 3 times every 28-day cycle
  Gemcitabine: Administer intravenously 3 times every 28-day cycle
- Gem/NP/Nivolumab/APX005M (0.1 mg/kg); Gem/NP/Nivolumab/APX005M (0.3 mg/kg): Gemcitabine+Nab-Paclitaxel+nivolumab+APX005M
  APX005M: Administer intravenously once every 28-day Cycle
  Nivolumab: Administer intravenously twice every 28-day cycle
  Nab-Paclitaxel: Administer intravenously on 3 times every 28-day cycle
  Gemcitabine: Administer intravenously 3 times every 28-day cycle
Arm/Group | Gem/NP/APX005M (0.1 mg/kg) | Gem/NP/APX005M (0.3 mg/kg) | Gem/NP/Nivolumab/APX005M (0.1 mg/kg) | Gem/NP/Nivolumab/APX005M (0.3 mg/kg)
Number analyzed (Participants) | 6 | 6 | 6 | 6
percentage of participants | 66.7 [22.28 to 95.67] | 33.3 [4.33 to 77.72] | 66.7 [22.28 to 95.67] | 66.7 [22.28 to 95.67]

4. Secondary Outcome: Duration of Response (DOR): DLT-Evaluable Population
Description: DOR was the time from the first tumor assessment demonstrating response until the date of radiographic disease progression. DOR and the CIs were estimated using the Kaplan-Meier method.
Time Frame: as for outcome 3
Population: Patients in the DLT-Evaluable Population (defined as all Phase 1b patients who received at least 2 doses of NP, at least 2 doses of Gem, and 1 dose of APX005M during Cycle 1) and who achieved a Partial Response or Complete Response.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Gem/NP/Nivolumab/APX005M (0.1 mg/kg): Gemcitabine+Nab-Paclitaxel+nivolumab+APX005M (0.1 mg/kg)
  APX005M: Administer intravenously once every 28-day Cycle
  Nivolumab: Administer intravenously twice every 28-day cycle
  Nab-Paclitaxel: Administer intravenously on 3 times every 28-day cycle
  Gemcitabine: Administer intravenously 3 times every 28-day cycle
Arm/Group | Gem/NP/APX005M (0.1 mg/kg) | Gem/NP/APX005M (0.3 mg/kg) | Gem/NP/Nivolumab/APX005M (0.1 mg/kg) | Gem/NP/Nivolumab/APX005M (0.3 mg/kg)
Number analyzed (Participants) | 4 | 2 | 4 | 4
months | 15.51 [1.54 to NA] — Some confidence limits are not estimable due to small sample sizes and censoring | 7.03 [6.01 to NA] — Some confidence limits are not estimable due to small sample sizes and censoring | 9.07 [NA to NA] — Some confidence limits are not estimable due to small sample sizes and censoring | 10.35 [5.32 to NA] — Some confidence limits are not estimable due to small sample sizes and censoring

5. Secondary Outcome: Disease Control Rate (DCR)
Description: Phase 2 Secondary Efficacy Outcome. Disease Control Rate is defined as the proportion of participants who had a best overall response of Complete Response (CR), Partial Response (PR), or Stable Disease (SD) as defined by RECIST v1.1.
Time Frame: Initiation of study drug through radiographic progression or initiation of new anti-cancer therapy with a maximum exposure of 24.2 months.
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Gem/NP/Nivolumab | Gem/NP/APX005M (0.3 mg/kg) | Gem/NP/Nivolumab/APX005M (0.3 mg/kg)
Number analyzed (Participants) | 34 | 36 | 35
percentage of participants | 73.5 [55.64 to 87.12] | 77.8 [60.85 to 89.88] | 68.6 [50.71 to 83.15]

6. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as the time from treatment initiation until radiographic disease progression or death (whichever occurred first). PFS and the CIs were estimated using the Kaplan-Meier method.
Time Frame: Initiation of study drug through radiographic progression or death with a maximum exposure of 24.2 months.
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Gem/NP/Nivolumab | Gem/NP/APX005M (0.3 mg/kg) | Gem/NP/Nivolumab/APX005M (0.3 mg/kg)
Number analyzed (Participants) | 34 | 36 | 35
months | 6.37 [5.19 to 8.80] | 7.26 [5.36 to 9.23] | 6.74 [4.17 to 9.79]

7. Secondary Outcome: Objective Response Rate (ORR): Efficacy Population
Description: Phase 2 Secondary Efficacy Outcome. Overall Response Rate is defined as the proportion of participants who had a best overall response of Complete Response (CR) or Partial Response (PR) as defined by RECIST v1.1. Overall Response (OR) = CR + PR.
Time Frame: as for outcome 5
Population: The Efficacy Population is defined as (1) all patients who were randomized in Phase 2 and who received at least 1 dose of any study drug and (2) the 12 DLT-evaluable patients enrolled in Phase 1b at the recommended Phase 2 dose (Arms B2 and C2).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Gem/NP/Nivolumab | Gem/NP/APX005M (0.3 mg/kg) | Gem/NP/Nivolumab/APX005M (0.3 mg/kg)
Number analyzed (Participants) | 34 | 36 | 35
percentage of participants | 50 [32.43 to 67.57] | 33.3 [18.56 to 50.97] | 31.4 [16.85 to 49.29]

8. Secondary Outcome: Duration of Response (DOR): Efficacy Population
Description: as for outcome 4
Time Frame: as for outcome 5
Population: Patients in the Efficacy Population (defined as all patients who were randomized in Phase 2 and who received at least 1 dose of any study drug and the 12 DLT-Evaluable patients enrolled in Phase 1b at the recommended Phase 2 dose) and who achieved a Partial Response or Complete Response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Gem/NP/Nivolumab | Gem/NP/APX005M (0.3 mg/kg) | Gem/NP/Nivolumab/APX005M (0.3 mg/kg)
Number analyzed (Participants) | 17 | 12 | 11
months | 7.36 [2.10 to NA] — The upper confidence limit is not evaluable due to insufficient number of participants with events | 5.55 [3.75 to 7.95] | 7.88 [1.91 to NA] — The upper confidence limit is not evaluable due to insufficient number of participants with events

ADVERSE EVENTS:
Time Frame: Adverse events were reported until 100 days after the last dose of study drug had been administered with a maximum exposure of 34.3 months.
Description: Safety analysis was conducted on all Phase 1b and Phase 2 patients who received at least one dose of any study drug. For safety analyses, patients were grouped according to the study treatment actually received ('as treated'). Specifically, two phase 2 patients were randomly allocated to Gem/NP/Nivolumab/APX005M but only received doses of Gem, NP, and Nivolumab (that is, APX005M was not received); these two patients were grouped as Gem/NP/APX005M for safety analyses.
Arm/Group | Gem/NP/Nivolumab | Gem/NP/APX005M (0.1 mg/kg) | Gem/NP/APX005M (0.3 mg/kg) | Gem/NP/Nivolumab/APX005M (0.1 mg/kg) | Gem/NP/Nivolumab/APX005M (0.3 mg/kg)
All-Cause Mortality (participants affected / at risk) | 25/36 | 5/7 | 29/37 | 8/8 | 27/35
Serious Adverse Events (participants affected / at risk) | 18/36 | 4/7 | 22/37 | 6/8 | 20/35
Other Adverse Events (participants affected / at risk) | 36/36 | 7/7 | 36/37 | 8/8 | 35/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gem/NP/Nivolumab (N=36) | Gem/NP/APX005M (0.1 mg/kg) (N=7) | Gem/NP/APX005M (0.3 mg/kg) (N=37) | Gem/NP/Nivolumab/APX005M (0.1 mg/kg) (N=8) | Gem/NP/Nivolumab/APX005M (0.3 mg/kg) (N=35)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Bile duct obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cardiac failure (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Demyelinating polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Facial nerve disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Haemoptysis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
IIIrd nerve disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Immune-mediated pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Incorrect dose administered (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Liver abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mesenteric venous occlusion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pneumonia staphylococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pseudocellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Pyrexia (General disorders) | 2 (2) | 0 (0) | 2 (2) | 3 (3) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 3 (3)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toxic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Gem/NP/Nivolumab (N=36) | Gem/NP/APX005M (0.1 mg/kg) (N=7) | Gem/NP/APX005M (0.3 mg/kg) (N=37) | Gem/NP/Nivolumab/APX005M (0.1 mg/kg) (N=8) | Gem/NP/Nivolumab/APX005M (0.3 mg/kg) (N=35)
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 5 | 0 | 7 | 2 | 8
Abdominal pain (Gastrointestinal disorders) | 15 | 0 | 15 | 3 | 18
Abdominal pain lower (Gastrointestinal disorders) | 4 | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 7 | 0 | 4 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 4 | 1 | 0
Adjustment disorder with anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Adjustment disorder with depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 18 | 4 | 22 | 1 | 23
Alopecia (Skin and subcutaneous tissue disorders) | 14 | 4 | 17 | 3 | 12
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 2
Anaemia (Blood and lymphatic system disorders) | 22 | 7 | 22 | 4 | 18
Anal fistula (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 9 | 1 | 9 | 0 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 2 | 4 | 2 | 4
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 4
Aspartate aminotransferase increased (Investigations) | 19 | 4 | 25 | 2 | 21
Asthenia (General disorders) | 2 | 3 | 4 | 3 | 2
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 1 | 0
Autoimmune neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 2 | 8 | 0 | 8
Blood alkaline phosphatase increased (Investigations) | 9 | 1 | 16 | 1 | 14
Blood bilirubin increased (Investigations) | 6 | 2 | 7 | 2 | 12
Blood creatine phosphokinase increased (Investigations) | 2 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 5 | 0 | 4 | 3 | 4
Blood potassium decreased (Investigations) | 0 | 1 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Candida infection (Infections and infestations) | 2 | 0 | 2 | 0 | 0
Cellulitis (Infections and infestations) | 2 | 1 | 2 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 3
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 2
Chills (General disorders) | 6 | 5 | 30 | 6 | 27
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 2
Confusional state (Psychiatric disorders) | 0 | 0 | 2 | 0 | 5
Constipation (Gastrointestinal disorders) | 16 | 2 | 22 | 4 | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 15 | 1 | 12 | 2 | 14
Cystitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 5 | 7 | 2 | 11
Decreased appetite (Metabolism and nutrition disorders) | 22 | 3 | 21 | 3 | 15
Deep vein thrombosis (Vascular disorders) | 2 | 1 | 5 | 0 | 4
Defaecation urgency (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 9 | 1 | 8 | 3 | 9
Delirium (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 6 | 2 | 7 | 0 | 6
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 19 | 3 | 20 | 3 | 21
Diplopia (Eye disorders) | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 7 | 3 | 6 | 1 | 9
Dry eye (Eye disorders) | 2 | 0 | 0 | 0 | 2
Dry mouth (Gastrointestinal disorders) | 3 | 0 | 4 | 0 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Dysarthria (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 4 | 3 | 4 | 3 | 7
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 5 | 0 | 5
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 | 4 | 14 | 2 | 13
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1 | 3
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 2
Early satiety (General disorders) | 2 | 0 | 0 | 1 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 | 3 | 7 | 0 | 6
Eructation (Gastrointestinal disorders) | 4 | 0 | 2 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 3
Face oedema (General disorders) | 0 | 0 | 3 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 0 | 2 | 1 | 2
Fatigue (General disorders) | 27 | 7 | 29 | 5 | 29
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 3 | 0 | 0
Flatulence (Gastrointestinal disorders) | 2 | 0 | 3 | 2 | 4
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Flushing (Vascular disorders) | 0 | 0 | 6 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 | 1 | 0 | 0 | 4
Generalised oedema (General disorders) | 0 | 1 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 0 | 1 | 0 | 2 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 8 | 2 | 12 | 4 | 4
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0
Hot flush (Vascular disorders) | 2 | 0 | 0 | 0 | 2
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 3 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 1 | 3 | 0 | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 6 | 0 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 0 | 3 | 0 | 2
Hypertension (Vascular disorders) | 4 | 1 | 9 | 1 | 5
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 2
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 4 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 7 | 2 | 3 | 1 | 4
Hypocalcaemia (Metabolism and nutrition disorders) | 3 | 0 | 2 | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 3 | 6 | 2 | 9
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 1 | 2 | 1 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 1 | 12 | 1 | 9
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 0 | 4 | 1 | 3
Hypotension (Vascular disorders) | 8 | 3 | 11 | 3 | 12
Hypothyroidism (Endocrine disorders) | 2 | 1 | 0 | 0 | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 4 | 2 | 3
Incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 2
Influenza like illness (General disorders) | 2 | 0 | 6 | 1 | 2
Infusion related reaction (Injury, poisoning and procedural complications) | 2 | 1 | 4 | 1 | 5
Infusion site pain (General disorders) | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 7 | 2 | 10 | 2 | 3
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 3 | 0 | 3 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 4
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 6 | 1 | 9 | 3 | 6
Lymphoedema (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Malaise (General disorders) | 3 | 1 | 3 | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 2 | 0 | 0 | 1 | 0
Medical device site joint swelling (General disorders) | 0 | 1 | 0 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 1 | 2 | 1 | 0
Mucosal inflammation (General disorders) | 3 | 1 | 5 | 1 | 5
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 0 | 2 | 0 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 10 | 0 | 10
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 | 2 | 3 | 0 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 2 | 0 | 3 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 4
Nausea (Gastrointestinal disorders) | 26 | 6 | 33 | 5 | 29
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 10 | 6 | 17 | 4 | 9
Neutropenia (Blood and lymphatic system disorders) | 8 | 4 | 12 | 1 | 6
Neutrophil count decreased (Investigations) | 13 | 4 | 15 | 2 | 15
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 4 | 0 | 3
Ocular icterus (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 2
Oedema (General disorders) | 0 | 3 | 3 | 1 | 5
Oedema peripheral (General disorders) | 15 | 2 | 22 | 3 | 13
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Oral pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 3 | 0 | 4
Otitis media (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Pain (General disorders) | 3 | 1 | 2 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 0 | 3 | 2 | 6
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 2 | 0 | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2
Paraesthesia (Nervous system disorders) | 0 | 1 | 5 | 0 | 2
Paronychia (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 3 | 1 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 8 | 0 | 7 | 2 | 7
Peripheral swelling (General disorders) | 0 | 2 | 2 | 0 | 2
Platelet count decreased (Investigations) | 13 | 3 | 13 | 3 | 17
Platelet count increased (Investigations) | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 2 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 3
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 4 | 1 | 0
Presyncope (Nervous system disorders) | 4 | 2 | 2 | 0 | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 1 | 16 | 2 | 13
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 1 | 4
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 16 | 4 | 29 | 6 | 24
Rash (Skin and subcutaneous tissue disorders) | 17 | 4 | 11 | 4 | 17
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 | 1 | 5 | 1 | 2
Renal failure (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 7 | 0 | 4
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 3 | 0 | 0
Sinusitis (Infections and infestations) | 2 | 0 | 2 | 1 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2
Skin wound (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 3
Splenic vein thrombosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 5 | 1 | 2 | 0 | 5
Tachycardia (Cardiac disorders) | 2 | 0 | 4 | 0 | 6
Taste disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 9 | 2 | 11 | 2 | 15
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 2 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Septic shock (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 6 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 1 | 2
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 2
Urinary tract infection (Infections and infestations) | 4 | 2 | 0 | 0 | 3
Urinary tract pain (Renal and urinary disorders) | 0 | 0 | 2 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 5 | 0 | 9
Vision blurred (Eye disorders) | 2 | 2 | 0 | 1 | 5
Visual acuity reduced (Eye disorders) | 0 | 1 | 0 | 0 | 0
Vitiligo (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 14 | 3 | 23 | 3 | 20
Weight decreased (Investigations) | 11 | 1 | 4 | 3 | 4
Weight increased (Investigations) | 0 | 0 | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1 | 2
White blood cell count decreased (Investigations) | 10 | 1 | 7 | 1 | 6
Pancreas infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 3
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 2
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Trial Site and/or Co-Principal Investigators may publish or present Study Data and other results of the Study from the Trial Site individually upon the first to occur of: (i) twelve (12) months after conclusion, abandonment, or termination of the Study at all Affiliated Research Institutions, or (ii) after Parker Institute for Cancer Immunotherapy [PICI] confirms in writing there will not be a multi-site Study publication.

DOCUMENTS (2):
  • Study Protocol (2019-10-11): https://cdn.clinicaltrials.gov/large-docs/50/NCT03214250/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-14): https://cdn.clinicaltrials.gov/large-docs/50/NCT03214250/SAP_001.pdf